CLINICAL TRIAL: NCT03603678
Title: Randomized, Multi-center, Double-blind, Placebo-controlled, Group-comparison Study to Investigate Safety, Tolerability and Pharmacodynamics of BAY2253651 After Administration of a Single Nasal Dose in 60 Subjects With Obstructive Sleep Apnea and Open Exploratory Evaluation of Safety and Local Tolerability of Repeated Doses in Patients
Brief Title: Obstructive Sleep Apnea (OSA) Treated With a Potassium Channel Inhibitor
Acronym: SANDMAN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19038; 2017-001851-29 (EudraCT Number)
Record Dates: First submitted 2018-06-21; First posted 2018-07-27 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Obstructive sleep apnea; Potassium channel blocker; Polysomnography; PSG
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part A single dose BAY2253651 (Experimental): Single dose BAY2253651
  Interventions: Drug: BAY2253651
- Part A single dose Placebo (Placebo Comparator): Single dose matching placebo
  Interventions: Drug: Placebo
- Part B multiple dose BAY2253651 (Experimental): Multiple dose BAY2253651 on 5 consecutive nights
  Interventions: Drug: BAY2253651

INTERVENTIONS:
Drug: BAY2253651 — 100 µg (500 µg/ml * 200 µl) BAY2253651 intranasally
  Arms: Part A single dose BAY2253651; Part B multiple dose BAY2253651
Drug: Placebo — Matching Placebo dosing
  Arms: Part A single dose Placebo

SUMMARY:
The aim of this study in subjects with obstructive sleep apnea is to investigate pharmacodynamics, safety and tolerability after a single nasal administration of BAY2253651 and to evaluate first safety and tolerability of multiple dosing over 5 consecutive nights in OSA patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects need to be diagnosed with OSA (obstructive sleep apnea) but should be otherwise healthy at the discretion of the investigator.
* Patients must be pretreated with CPAP (continuous positive airway pressure) for OSA for at least 3 months before randomization.
* AHI of 15-50 per hour after 48 hours of CPAP withdrawal documented by baseline PSG (polysomnography, evaluated by the site staff) and at least 4 hours of total sleep time. (One retesting allowed).
* Female subjects must be of non-childbearing potential, i.e. post-menopausal (no menses for at least 1 year prior to randomization) or surgically sterile (tubal ligation, hysterectomy or bilateral oophorectomy)
* Men of reproductive potential together with their female partner(s) must agree to use at least two adequate contraception methods when sexually active. This applies for the time period between signing of the informed consent form and 3 months after the last administration of study drug.

Acceptable methods of contraception include, but are not limited to, (i) condoms (male or female) with or without a spermicidal agent; (ii) diaphragm or cervical cap with spermicide; (iii) intra-uterine device; (iv) hormone-based contraception

* Only Part B: Patients having completed Part A and had valid PSG after dosing in Part A.

Exclusion Criteria:

* Inability to comply with planned study procedures or to comply with study protocol requirements; this includes completing required data collection and attending required follow up study visits.
* Neck circumference above/equal 44 cm.
* Not predominantly obstructive sleep apnea evidenced by baseline PSG.
* Severely impaired breathing within two days prior to randomization (e.g. acute nasal congestion during upper airway infection).
* Subject with known allergies or hypersensitivities to the study drugs (active substances or excipients of the preparations). Known severe respiratory tract allergies e.g. allergic asthma.
* Intake of a nasal decongestant during the intervention time (48 hours before visit 1 until end of visit 2).
* Use of any topical medication containing local anesthetics for nose and throat within 7 days before first investigational medicinal product (IMP) administration.
* Participation in another trial with an investigational drug within 30 days or 5 half-lives of the investigational drug, whichever is longer before first application of study drug or concomitant participation in another clinical study with investigational medicinal product(s).
* Any other condition, which would make the subject unsuitable for this study and will not allow participation for the full planned study period (e.g. active malignancy or other condition limiting life expectancy to less than 12 months)
* Known history of severe heart failure (NYHA 3-4) or severe COPD (GOLD 3-4).
* Heavy smoking, i.e. more than 20 cigarettes per day and/or unable to stop smoking during the stay in the sleep laboratory.
* Suspicion of drug or alcohol abuse.
* Regular daily consumption of more than 1 L of xanthine-containing beverages.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2019-05-23 (Actual); Study Completion 2019-09-02 (Actual)

PRIMARY OUTCOMES:
Rate of responders, defined by reduction of apnoea-hypopnoea-index (AHI) from baseline by ≥ 50% | 2 days

SECONDARY OUTCOMES:
Incidence of treatment emergent adverse events (TEAEs) | Up to 7 days
Severity of treatment emergent adverse events (TEAEs) | Up to 7 days

CONTACTS AND LOCATIONS:
Locations (2):
- University Hospital Zürich, Zurich, Switzerland
- Oxford University Hospitals, Oxford, United Kingdom

REFERENCES:
- [Derived] Gaisl T, Turnbull CD, Weimann G, Unger S, Finger R, Xing C, Cistulli PA, West S, Chiang AKI, Eckert DJ, Stradling JR, Kohler M. BAY 2253651 for the treatment of obstructive sleep apnoea: a multicentre, double-blind, randomised controlled trial (SANDMAN). Eur Respir J. 2021 Nov 18;58(5):2101937. doi: 10.1183/13993003.01937-2021. Print 2021 Nov. PMID 34531274